CLINICAL TRIAL: NCT05921656
Title: Construction and Evaluation of Airway Leakage Risk Model of Patients With Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Honglei Wu, the investigators, Affiliated Hospital of Nantong University
Other Study IDs: 2021-K062-01
Record Dates: First submitted 2023-04-11; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Mechanical Ventilation
MeSH Terms: interventions — Facility Design and Construction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Construction and evaluation of airway leakage risk model of patients with endotracheal tube — 1. Conduct statistical analysis on general information, respiratory data, tracheal catheter data, and cross-sectional area of the patient's airway to clarify the current status of airway leakage and related influencing factors.
  2. Based on multivariate logistic regression, a line chart prediction model for predicting the risk of airway leakage in patients with tracheal catheters is constructed. The clinical efficacy of the prediction model is evaluated by using the area under the ROC curve, the Calibration scatter plot, and the DCA decision line, respectively, to assess its discrimination, calibration, and clinical practicality.

SUMMARY:
There are two cases in which the cross-sectional area of the tracheal catheter balloon does not match the cross-sectional area of the patient's airway. If the area of the tracheal catheter balloon is smaller than the cross-sectional area of the patient's airway, the pressure in the balloon reaches 30 cmH2O, and the airway cannot be completely sealed; This will increase the risk of VAP. If the area of the tracheal catheter balloon is significantly larger than the cross-sectional area of the patient's airway, and the pressure in the balloon reaches 30 cmH2O, the airway cannot be effectively sealed; The formation of wrinkles around the airbag also increases the risk of VAP in patients. Therefore, the purpose of this study is to build a risk model of airway leakage of patients' endotracheal tubes, which provides an accurate and objective assessment tool for medical staff, so that medical staff can select the endotracheal tubes purposefully and with emphasis from the beginning of the patients' endotracheal tubes, and reduce the airway leakage or airway mucosal damage of the endotracheal tubes.

DETAILED DESCRIPTION:
Admission number, department, name, gender, height, and weight are obtained through the hospital's electronic medical record management system。 Tidal volume (set Tidal volume), airway peak pressure (real-time data on the ventilator screen), data collection is synchronized with the minimum cuff pressure measurement when the airway is closed.

ELIGIBILITY:
Inclusion Criteria:

Invasive mechanical ventilation; Chest CT imaging examination within 1 year;

Exclusion Criteria:

Patients with pneumothorax Acute respiratory distress syndrome; Chronic Obstructive Pulmonary Disease; Multiple organ dysfunction.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators selected mechanical ventilation patients admitted to the Extracardiac and Respiratory Care Units of Nantong University Affiliated Hospital from September 2021 to September 2022 who underwent cardiac, pulmonary, esophageal surgery, and other procedures as the research subjects.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Patient airway area | Within 1 year
  Firstly, confirm the front position of the tracheal catheter through chest X-ray, and then manually sketch the area of interest along the outer wall of the airway using Computed Tomography to calculate the area.

SECONDARY OUTCOMES:
Measure the minimum cuff pressure | 1min
  The specific method is as follows: the patient takes a 30 ° semi recumbent position, puts a Stethoscope on the throat of the patient's trachea, inflates air into the trachea tube cuff until the air leakage sound just disappears, at this time, the value displayed by the cuff pressure gauge is the minimum cuff pressure when the airway is closed

CONTACTS AND LOCATIONS:
Overall Officials: HongLei wu, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

REFERENCES:
- [Result] Selman Y, Arciniegas R, Sabra JM, Ferreira TD, Arnold DJ. Accuracy of the minimal leak test for endotracheal cuff pressure monitoring. Laryngoscope. 2020 Jul;130(7):1646-1650. doi: 10.1002/lary.28328. Epub 2019 Oct 8. PMID 31593330